CLINICAL TRIAL: NCT03810989
Title: Using of the Skin as a Third Spare Kidney for Patients With Chronic Renal Failure
Brief Title: Dermodialysis as Adjuvant Therapy in Renal Failure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Yasser Abd Elmawgood Fysal Ibrahim, assistant lecturer, Assiut University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: skin as third kidney
Record Dates: First submitted 2019-01-17; First posted 2019-01-22 (Actual); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Chronic Renal Failure
Keywords: dermodialysis
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Intervention Model Description: the same groups of patients will be used for the experimental and control groups (self controlled study or time series study).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- infra-red sauna (Experimental): During the intervention phase, the patient will be dialysed twice weekly on Saturday and Wednesday. During the in-between three days, the patients will be subjected to an intervention as the following :- three session of infra-red sauna of 15 minutes duration separated by ten minutes rest outside the sauna.
  Interventions: Device: infra-red sauna
- argometer and treadmill (Experimental): During the intervention phase, the patient will be dialysed twice weekly on Saturday and Wednesday. During the in-between three days, the patients will be subjected to an intervention as the following :- three session of physical exercise (by treadmill and argometer) of 20-30 minutes duration separated by 10 minutes rest.
  Interventions: Device: argometer and treadmill
- combination of sauna and hot bath (Experimental): During the intervention phase, the patient will be dialysed twice weekly on Saturday and Wednesday. During the in-between three days, the patients will be subjected to an intervention as the following :- three session of infra-red sauna as the first group then the patients will be immersed up to neck for one hour in water at 37-43 C.
  Interventions: Device: combination of sauna and hot bath
- combination of sauna and hot bath in CKD (Experimental): During the ﬁrst month (control phase), S Cr, BUN, serum K and serum phosphorus will be measured weekly and the mean will be calculated. During the next two months (intervention phase) the patient will be subjected to three session of sauna of 15 minutes duration separated by ten minutes rest outside the sauna then the patients will be immersed up to neck for one hour in water at 37 -43 C .
  Interventions: Device: combination of sauna and hot bath

INTERVENTIONS:
Device: infra-red sauna — During the intervention phase, the ESRD patients twill be subjected to a method of stimulation of sweating as the following :- three session of infra-red sauna of 15 minutes duration separated by ten minutes rest outside the sauna.
  Arms: infra-red sauna
Device: argometer and treadmill — During the intervention phase, the ESRD patients twill be subjected to a method of stimulation of sweating as the following :- three session of physical exercise (by treadmill and argometer) of 20-30 minutes duration separated by 10 minutes rest.
  Arms: argometer and treadmill
Device: combination of sauna and hot bath — During the intervention phase, the ESRD patients twill be subjected to a method of stimulation of sweating as the following :- three session of infra-red sauna as the first group then the patients will be immersed up to neck for one hour in water at 37-43 C.
  Arms: combination of sauna and hot bath; combination of sauna and hot bath in CKD

SUMMARY:
Using sweat as the vehicle for removing molecules normally excreted in the urine(dermodialysis) was identified some decades ago.The study will include 66 ESRD patients and 20 CKD stage 5 patients not on dialysis who met inclusion and exclusion criteria. The ESRD patients will be divided into three groups and will be subjected to different modalities of stimulation of sweating like infra-red sauna , physical exercise and hot bath. The study will be conducted over a period of three months. During the ﬁrst month, patients were dialyzed as usual (control phase).During the next two months ,the participants will be dialysed twice weekly in addition to dermodialysis. S Cr, BUN, serum K and serum phosphorus will be measured weekly immediately before the last dialysis session during the control and intervention phases. The mean of this investigations during each phase will be calculated . The investigators will compare the mean of this investigations during control phase with the mean during the intervention phase to evaluate the effectiveness of dermodialysis as adjuvant therapy for ESRD patients.The patients not on dialysis will subjected to infra-red sauna and hot bath.The investigators also will compare the means of S Cr, BUN, serum K and serum phosphorus during both control and intervention phases like the ESRD patients.

DETAILED DESCRIPTION:
Although dialysis has been considered as a life-saving treatment for end stage renal disease (ESRD) patients, many ESRD patients in developing countries don't have access to dialysis facilities . Using sweat as the vehicle for removing molecules normally excreted in the urine(dermodialysis) was identified some decades ago. Sweat fluid mainly contains sodium chloride, potassium, urea, ammonia, uric acid, and creatinine. The mean sweat fluid urea concentration could reach 5.5 to 50 times the serum concentration . In particular, urea concentrations in human sweat are persistently elevated in uremic patients . The 24-hour urinary urea excretion in summer was as much as one-quarter of the quantity in winter in uremic patients, indicating the compensatory urea excretion in sweat gland fluid .This high level of urea and other toxic molecules crystallize out and deposit visibly on the skin when the water of the sweat evaporates off ('uremic frost') .Sweat K concentration was significantly higher in ESRD patients . Pruijm, El-Housseini et al reported that stimulated sweating can be an effective way to reduce intradialytic weight gain(IDWG) in hemodialysis( HD)patients. These findings indicated that dermodialysis can be used to delay the requirement for and to reduce the frequency of dialysis and to improve the quality of lives of ESRD patients especially in the developing World where economic and technical support barriers to the provision of dialysis are present.

Sweating can be stimulated by many methods like physical exercise ,saunas and drugs like pilocarpine. Traditional dry saunas use temperatures as high as 185 to 195 degrees F, which is too much for some patients to tolerate. Infrared saunas use a much lower temperature (120 to 150 degrees F). However, because the heat of infrared saunas travels much deeper into the body, they are able to cause a more vigorous sweat at lower temperature. Infrared sauna has many benefits like normalizing blood pressure , treating congestive heart failure, weight loss and relieving of chronic pain.

Head out water immersion was used many times in ESRD patients. Pruijm, El-Housseini et al concluded that immersion in hot bath (temperature 37-43C) was effective method of stimulating sweating and reducing IDWG. Intradialytic hypotension could be prevented by water immersion.

Primary objective:- Evaluation of feasibility of dermodialysis as adjuvant replacement therapy for ESRD patients to decrease the cost of dialysis facilities (one third of the total cost).

Secondary objectives:-

1. Improve uremic pruritus.
2. Better control of blood pressure.
3. Decrease interdialytic weight gain.
4. Comparing the effectiveness of infra-red sauna, exercise and combination of infra-red sauna and head out water immersion as modality of dermodialysis The study will include 66 ESRD patients and 20 CKD stage 5 patients not on dialysis who met inclusion and exclusion criteria. The ESRD patients will be subdivided into three group, each group will include 22 patients .Each group will be subjected to Detailed history and Careful examination. The study will be conducted over a period of three months(for each patient). During the ﬁrst month, patients will be dialyzed as usual (control phase). Detailed information on blood pressure, interdialytic weight gain (IDWG), and dialysis prescription will be recorded. S Cr, BUN, serum K and serum phosphorus will be measured weekly immediately before the last dialysis session for one month and the mean will be calculated. During the next two months the patient will be dialysed twice weekly on Saturday and Wednesday. during the in-between three days(Sunday, Monday and Tuesday) the three groups subjected to intervention as the following :- Group 1:-three session of infra-red sauna of 15 minutes duration separated by ten minutes rest outside the sauna.

Group 2:-three session of physical exercise of 20-30 minutes duration separated by 10 minutes rest.

Group 3:-three session of infra-red sauna as the first group then the patients will be immersed up to neck for one hour in water at 37-43 C.

Detailed information on IDWG, blood pressure, any improvement in uremic pruritus will be recorded. Body temperature before and after the intervention will be measured and recorded. Assessment of uremic pruritus according to verbal rating scale (VRS) which divided into four level:-0=no symptom, 1=mild, 2= moderate, 3=sever or intense symptom. Dialysis prescription and diet will be fixed as possible to be similar to the control phase.

S Cr, BUN, serum K and serum phosphorus will be measured weekly immediately before the last dialysis session (Wednesday) for two months and the mean will be calculated. The patients will be admitted in internal medicine department in the dialysis free period to be under close observation. Dialysis will be done if there is urgent indication in the dialysis free days.

The CKD group :- The patients will be subjected to Detailed history and Careful examination. The study will be conducted over a period of three months. During the ﬁrst month (control phase), S Cr, BUN, serum K and serum phosphorus will be measured weekly and the mean will be calculated. During the next two months the patient will be subjected to three session of sauna of 15 minutes duration separated by ten minutes rest outside the sauna then the patients will be immersed up to neck for one hour in water at 37 -43 C . Body temperature before and after the intervention will be measured and recorded. During the intervention phase, S Cr, BUN, serum K and serum phosphorus will be measured weekly and the mean will be calculated. During the period of rest the patients will consume sufficient amount of water to avoid dehydration .Blood pressure will be monitored and recorded. Dialysis will be done if there is urgent indication or standard indication for dialysis according to KDOQI guide lines 2015.

ELIGIBILITY:
Inclusion Criteria:

* A-chronic renal failure groups:-

  1. Patients with chronic renal failure on regular haemodialysis three times a week.
  2. starting regular haemodialysis at least 6 months before the beginning of the study.
  3. Ability to perform physical exercise in argometer and treadmill arm.
* B-chronic kidney disease(CKD) group:

  * 1- CKD stage 5 (eGFR 10-15ml /min calculated by EPI equation).

    2-Not on dialysis.

    3-Without uremic symptoms nor standard indication for dialysis according to KDOQI guide lines.

Exclusion Criteria:

* A-ESRD groups:-

  1. Having temporary or tunneled catheter as modality of vascular access.
  2. History of cerebrovascular accidents.
  3. History of advanced cardiac disease (heart failure, recent acute coronary syndrome, and cardiac arrhythmia).
  4. Active skin lesion
  5. large ultrafiltration volume per session(>2 Litter)
  6. Patients with dry skin.

-B-chronic kidney disease (CKD) group:-

1. Diabetes mellitus .
2. History of advanced heart failure, advanced liver cirrhosis, respiratory failure, and malignancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2019-06-01 (Estimated); Primary Completion 2020-06-01 (Estimated); Study Completion 2020-09-01 (Estimated)

PRIMARY OUTCOMES:
change in the mean of BUN, serum Cr, serum k and serum phosphorus . | 3months
  S Cr, BUN, serum K and serum phosphorus will be measured weekly immediately before the last dialysis session during the control and intervention phases. The mean of this investigations during each phase will be calculated .The investigators will compare the mean of this investigations during control phase with the mean during the intervention phase to evaluate the effectiveness of dermodialysis as adjuvant therapy for ESRD patients.
change in interdialytic weight gain(IDWG) | 3months
  interdialytic weight gain(IDWG)=weight of the patients before the dialysis session minus his weight immediately after the previous session. The mean of IDWG will be calculated during both the control and intervention phases ,then The investigators will compare both means.

SECONDARY OUTCOMES:
The effect on uremic pruritus | 3 months
  Assessment of uremic pruritus according to verbal rating scale (VRS) during both control and intervention phases . Verbal rating scale (VRS)which divided into four level:-0=no symptom, 1=mild, 2= moderate, 3=sever or intense symptom.the investigators will compare the severity of uremic pruritus in the two phases.

CONTACTS AND LOCATIONS:
Overall Officials: Ashraf Elshazly, professor, Study Director — Assiut University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Yosipovitch G, Reis J, Tur E, Blau H, Harell D, Morduchowicz G, Boner G. Sweat electrolytes in patients with advanced renal failure. J Lab Clin Med. 1994 Dec;124(6):808-12. PMID 7798794
- [Background] Mohan D, Railey M. Uremic frost. Kidney Int. 2012 Jun;81(11):1153. doi: 10.1038/ki.2012.70. No abstract available. PMID 22584601
- [Background] Huang CT, Chen ML, Huang LL, Mao IF. Uric acid and urea in human sweat. Chin J Physiol. 2002 Sep 30;45(3):109-15. PMID 12817713
- [Background] al-Tamer YY, Hadi EA, al-Badrani II. Sweat urea, uric acid and creatinine concentrations in uraemic patients. Urol Res. 1997;25(5):337-40. doi: 10.1007/BF01294662. PMID 9373914
- [Background] Barsoum RS. Chronic kidney disease in the developing world. N Engl J Med. 2006 Mar 9;354(10):997-9. doi: 10.1056/NEJMp058318. No abstract available. PMID 16525136
- [Background] El Nahas M. The global challenge of chronic kidney disease. Kidney Int. 2005 Dec;68(6):2918-29. doi: 10.1111/j.1523-1755.2005.00774.x. No abstract available. PMID 16316385
- [Background] Modi GK, Jha V. The incidence of end-stage renal disease in India: a population-based study. Kidney Int. 2006 Dec;70(12):2131-3. doi: 10.1038/sj.ki.5001958. Epub 2006 Oct 25. PMID 17063176
- [Result] Snyder D, Merrill JP. Sauna baths in the treatment of chronic renal failure. Trans Am Soc Artif Intern Organs. 1966;12:188-92. No abstract available. PMID 5960700
- [Result] Lacher JW, Schrier RW. Sweating treatment for chronic renal failure. Nephron. 1978;21(5):255-9. doi: 10.1159/000181401. PMID 714199
- [Result] Vance DJ. Dermodialysis-Could sweating treatments for chronic renal failure substantially and feasibly improve outcomes in developing and even developed world contexts?
- [Result] Pruijm M, El-Housseini Y, Mahfoudh H, Jarraya F, Hachicha J, Teta D, Burnier M. Stimulated sweating as a therapy to reduce interdialytic weight gain and improve potassium balance in chronic hemodialysis patients: a pilot study. Hemodial Int. 2013 Apr;17(2):240-8. doi: 10.1111/j.1542-4758.2012.00751.x. Epub 2012 Sep 26. PMID 23013432
- [Result] Doenyas-Barak K, Garra N, Beberashvili I, Efrati S. Immersion-enhanced fluid redistribution can prevent intradialytic hypotension: A prospective, randomized, crossover clinical trial. Hemodial Int. 2018 Jul;22(3):377-382. doi: 10.1111/hdi.12634. Epub 2018 Feb 13. PMID 29436152
- [Result] Beever R. Far-infrared saunas for treatment of cardiovascular risk factors: summary of published evidence. Can Fam Physician. 2009 Jul;55(7):691-6. PMID 19602651